CLINICAL TRIAL: NCT06833814
Title: DOSE Trial: Optimal Dose of Oral Corticosteroids to Treat Asthma Exacerbations: A Parallel, Randomized Controlled Pilot Study
Brief Title: DOSE Trial: Optimal Dose of Oral Corticosteroids to Treat Asthma Exacerbations
Acronym: DOSE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Andréanne Côté (Other)
Responsible Party: Sponsor-Investigator, Andréanne Côté, Respirologist-intensivist, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-4274
Record Dates: First submitted 2025-02-07; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Asthma Exacerbations
Keywords: asthma exacerbation; prednisone; randomized controlled trial
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Small-dose short-course (Experimental): 3 days of 50 mg of prednisone followed by 7 days of placebo
  Interventions: Drug: Prednisone
- Usual care (Active Comparator): 3 days of 50 mg of prednisone and 4 days of 25 mg of prednisone followed by 3 days of placebo
  Interventions: Drug: Prednisone
- High-dose long-course (Active Comparator): 5 days of 50 mg of prednisone and 5 days of 25 mg of prednisone
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Either 150 mg over 3 days or 250 mg over 7 days or 350 mg over 10 days

SUMMARY:
Patients with severe asthma frequently experience exacerbations of their disease. The heterogeneity of asthma exacerbations represents a major challenge for patients and healthcare providers, making treatment difficult. Current guidelines recommend varying doses of short-term oral corticosteroids (OCS) as first-line treatment for asthma exacerbations. However, studies supporting the optimal dose of OCS to treat asthma exacerbations are rare.

This study aims to evaluate the feasibility, acceptability, and safety of a randomized clinical trial with different OCS regimens for patients and physicians. Additionally, evaluate the success rate of different OCS dosages to support power calculations for a non-inferiority trial.

In this pilot, parallel, randomized, controlled study, patients with severe asthma exacerbation, considered to require treatment with OCS according to physician judgment after a complete evaluation will be randomized to 1) 3 days of 50 mg prednisone followed by 7 days of placebo, 2) 3 days of 50 mg prednisone and 4 days of 25 mg prednisone followed by 3 days of placebo, or 3) 5 days of 50 mg prednisone and 5 days of 25 mg prednisone. Randomized patients will be assessed for daily symptoms and overall perception of well-being, in addition to asthma control, quality of life as well as additional medical visits. Lung function and inflammation will also be measured. Feasibility and acceptability will be defined by a participation rate >80%, while safety will be defined as an increase in OCS doses in <20% of patients in one arm or an emergency room visit in <10% of patients in one arm. Success will be defined as no increased or prolonged doses of OCS, no re-consultation for OCS or escalation to antibiotics, reduction of symptoms, and return of lung function to >80% of its optimal level.

In addition to determining the feasibility and safety of different OCS regimens to treat asthma exacerbations, this trial will help us determine the optimal design for a randomized clinical trial using different OCS regimens. The exacerbation clinic is already operational with 4 to 5 patients/week assessed and treated. We have all the resources on site to carry out this project.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers
* 18 years of age or older
* Assessed for a severe asthma exacerbation
* Being prescribed OCS for the management of their exacerbation
* Able to comprehend and follow all required study procedures
* Able to understand and give written informed consent and have signed a written informed consent form (ICF) approved by the REB

Exclusion Criteria:

* For females, are pregnant, or lactating
* Respiratory comorbidities other than asthma, including bronchiectasis (non-CF) or asthma-COPD overlap (ACO)
* FEV1 <40% of personal best or <1 Li
* OCS-dependent
* Asthma exacerbation in the 4 weeks preceding the study visit
* Concomitant disease, health condition, and/or lifestyle activities that could interfere with the conduct of the study, or for which the treatment might interfere with the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study, including, but not limited to, cancer, alcoholism, drug dependency or abuse, or psychiatric disease. These include, but are not restricted to: heart failure, previous bipolar decompensation with prednisone, severe blood hypertension, uncontrolled diabetes, pneumonia.
* Unwilling or unable to comply with the study protocol for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02-17 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate | 9 months
  Period of time needed to recruit the total number of subjects.
Acceptability | 9 months
  Acceptability for subjects will be defined by the proportion of subjects agreeing to the study whereas acceptability for physicians will be defined by the proportion of subjects for whom the physicians prescribe OCS and is willing to enroll them in the study.

SECONDARY OUTCOMES:
Safety outcome: emergency room visits | 14 days
  Did the participant go to the emergency room visit between day of exacerbation and day 14.
Safety outcomes: Hospitalization | 14 days
  Was the patient hospitalized between day of exacerbation and day 14?
Safety outcomes: Unscheduled medical visits | 14 days
  Did the participant go for an unscheduled medical visit between day of exacerbation and day 14?
Safety outcomes: increased or prolonged OCS dose | 14 days
  Has the participant had to increase or prolong his OCS dose?
Safety outcomes: New or increase antibiotics | 14 days
  Was the participant prescribed new antibiotics treatment or had to increase antibiotics between day of exacerbation and day 14?

OTHER OUTCOMES:
Success rate | 14 days
  Success parameters will include increased or prolonged OCS dose, re consultation for OCS, new, increased or prolonged antibiotics, change in ACQ6 score between baseline and 14 days, and change in FEV1 between baseline and 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Andréanne Côté, MD-MSc, Principal Investigator — IUCPQ-UL

IPD SHARING:
Plan to Share IPD: Undecided